CLINICAL TRIAL: NCT00570609
Title: CPR Training in 7th Grade Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marna Rayl Greenberg (Other)
Responsible Party: Sponsor-Investigator, Marna Rayl Greenberg, Director of Emergency Medicine Research, Lehigh Valley Hospital
Organization: Lehigh Valley Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2-20070909
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Atherosclerosis; Prevention of Heart Disease
Keywords: CPR
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CPR Anytime (Experimental): Participants will be asked to complete the program with their parent(s)/legal guardian(s) and encouraged to include other friends and family members in the program
  Interventions: Other: CPR Anytime education

INTERVENTIONS:
Other: CPR Anytime education — After consent, participants will be asked to complete the 22 minute DVD CPR Anytime program with their parent(s)/legal guardian(s) and encouraged to include other friends and family members in the program

SUMMARY:
This is a prospective study of 7th grade students participating in the CPR Anytime® program. After consent, participants will be asked to complete the program with their parent(s)/legal guardian(s) and encouraged to include other friends and family members in the program. After completing the program, the participant and their parent(s) will be evaluated for adequacy of chest compressions/CPR. The student participants will be evaluated again at 6 months for adequacy of chest compressions/CPR

Objectives:

1. To evaluate 7th grade students for adequacy of CPR and chest compressions after completing a take home CPR course
2. To evaluate the multiplier effect of students training in CPR with their parents/family members using a take home CPR instructional kit
3. To evaluate the participating parent for adequacy of CPR and chest compressions after completing a take home CPR course

Research Hypothesis:

1. 7th grade students can be trained, using CPR Anytime®, to perform adequate chest compressions/CPR and their skills will be maintained at 6 months
2. As part of the multiplier effect, an additional 1.5 family members per participant will be trained to perform adequate chest compressions/CPR

DETAILED DESCRIPTION:
Participants will be selected from Salisbury and Swain schools. Parents and students from the participating schools will be invited by the school to an educational assembly in the fall of 2007. The material covered in the assembly will include issues of heart health and the importance of CPR. At the conclusion of the educational session, a description of the proposed study will be presented. The description will include details of the study and consent process. The consent and assent will be explained in detail to the prospective participants. The description of the study and consent/assent process will be delivered by one of the study investigators/coordinators. Details of the consent/assent will also be given to the prospective participants in a written format

For those potential participants unable to attend the assembly, consent and assent forms will be sent home with the student. Description of the project and explanation of the assent/consent process will be included. The potential participants will be encouraged to contact a study team member should they have any questions relating to the project or assent/consent process. Potential participants will be asked to return to the school on the projected date of CPR evaluations. The study team members will have the opportunity during this meeting to explain the study procedures as well as obtaining assent/consent.

After obtaining consent/assent, participants will be given a CPR Anytime kit and asked to complete the training at home with their parent(s)/guardian(s). They will also be encouraged to invite other family members and friends to participate with them in the training. All students in the 7th grade whether they participate in the study or not at the respective schools will receive a CPR Anytime kit.

The kit consists of a portable inflatable CPR training mannequin, a CPR training booklet, a 22 minute training DVD, and cleaning towelettes.

After completing the training, the student and parent participants will be evaluated for quality of CPR/chest compressions by a trained CPR instructor. The evaluation will be done on an individual basis not as a group. If remediation is required, it will take place at the time of the evaluation. The evaluation will be done at the school. The student participant will return at approximately months for reevaluation by the CPR instructor.

The student and parent participants will be asked to complete a survey at the time of initial training. The student participant will be asked to complete a follow up survey at the 3 month follow up

The data collected will be entered into a database. Each participant will be given a study identification number and data will be entered into the database using that number. The surveys will be anonymous. The participants will be identified by name on the CPR evaluations. Those families who receive the CPR Anytime kit but do not participate in the research study for testing will be surveyed to see how they used the kit in their home.

All hard copies (surveys and evaluation forms ) will be destroyed immediately after the data has been entered into the database. Access to the data will be limited to the PI and study coordinators. The hard copies and database will be stored in the research office and the office will be locked when not in use.

ELIGIBILITY:
Inclusion Criteria:

1. Participants
2. Access to home DVD player
3. Participants must be able to read, speak and understand English

Exclusion Criteria:Exclusion Criteria:

1. Lack of functioning home DVD player
2. Physical limitation to the ability to perform CPR/Chest compressions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
As tested by a CPR instructor, 7th grade students will be evaluated for performance of adequate chest compressions/CPR initially and at at 6 months after training with CPR Anytime®, | 6 months

SECONDARY OUTCOMES:
As part of the multiplier effect, an additional 1.5 family members per participant will be expected to be trained to perform adequate chest compressions/CPR | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marna R Greenberg, D.O., MPH, Principal Investigator — LVH
Locations (1):
- Salisbury Middle School, Allentown, Pennsylvania, United States